CLINICAL TRIAL: NCT06590402
Title: A Pilot Study Comparing Anterior Femoral Cutaneous Nerve Blocks to Adductor Canal Blocks in Pediatric Ambulatory Knee Surgeries
Brief Title: Anterior Femoral and Adductor Canal Nerve Blocks in Peds Knees
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2024-0582
Record Dates: First submitted 2024-08-06; First posted 2024-09-19 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Medial Patellofemoral Ligament Reconstruction
MeSH Terms: interventions — Bupivacaine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: A double-blinded pilot parallel group-randomized trial (GRT), subjects are enrolled and randomized based on their condition, and there is no cross-over of the groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of the patient/parent or guardian and research staff collecting data will be maintained via the "SNOSE" technique (Sequentially Numbered Opaque Sealed Envelope), whereby prior to study start, a research staff member not otherwise involved in the study will prepare envelopes with the randomization written on the card and secured in the envelopes, and the study ID number written outside the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Anterior Cruciate Ligament (ACL) surgeries (Experimental): Pediatric subjects who underwent a Anterior Cruciate Ligament (ACL) surgery and are randomized to receive either the adductor canal block (ACB) or the anterior femoral cutaneous nerve block (AFCNB).
  Interventions: Drug: Bupivacaine, Dexamethasone in Adductor Canal Block; Drug: Bupivacaine, Dexamethasone in Anterior Femoral Cutaneous Nerve Block
- Medial Patellofemoral Ligament (MPFL) surgeries (Experimental): Pediatric subjects who underwent a Medial Patellofemoral Ligament (MPFL) surgery and are randomized to receive either the adductor canal block (ACB) or the anterior femoral cutaneous nerve block (AFCNB).
  Interventions: Drug: Bupivacaine, Dexamethasone in Adductor Canal Block; Drug: Bupivacaine, Dexamethasone in Anterior Femoral Cutaneous Nerve Block

INTERVENTIONS:
Drug: Bupivacaine, Dexamethasone in Adductor Canal Block — 0.25% 15-20ml bupivacaine (local anesthestic) delivered as part of the adductor canal block with 2 mg preservative-free dexamethasone (corticosteroid) delivered as part of the adductor canal block
  Other Names: Adductor Canal Block (ACB)
Drug: Bupivacaine, Dexamethasone in Anterior Femoral Cutaneous Nerve Block — 10 ml of 0.25% bupivacaine (local anesthetic) delivered as part of the anterior femoral cutaneous nerve block with 2 mg preservative-free dexamethasone (corticosteroid) delivered as part of the anterior femoral cutaneous nerve block
  Other Names: Anterior Femoral Cutaneous Nerve Block (AFCNB)

SUMMARY:
The goal of this pilot clinical trial is to compare anterior femoral cutaneous nerve block (AFCN) to adductor canal block ACB) for pediatric patients undergoing either anterior cruciate ligament (ACL) or medial patellofemoral ligament (MPFL). The aims of this trial are:

* To measure postoperative functional outcomes in patients who received AFCNB vs. ACB.
* To calculate postoperative opioid requirements in pediatric knee surgeries that received AFCNB vs. ACB.
* To calculate pain intensity levels at rest and with ambulation in patients who received AFCNB vs. ACB.
* To quantify sensory deficits in patients who received AFCNB vs. ACB.
* To assess patient-reported outcome measures (e.g., pain expectation scale, pain management satisfaction, PROMIS Pediatric Short Form v1.0 - Physical Activity, PROMIS Scale v1.2 - Global Health) in patients 8-18 years of age who received AFCNB vs. ACB.

Subjects undergoing ACL procedures will be compared between those who received the adductor canal block to those who received the anterior femoral cutaneous nerve block. The researchers will also compare individuals who underwent MPFL procedures and received an anterior femoral cutaneous nerve block with those who received the adductor canal block.

Participants will:

* Be randomized to receive either the AFCNB or ACB in addition to standard of care analgesia.
* Maintain a patient diary to document daily pain meds/pain scores
* Complete follow up surveys/questionnaires via telephone and during their office visits with surgeons.

DETAILED DESCRIPTION:
There is scant literature on the efficacy of peripheral nerve blocks or the comparative effectiveness of anesthesia and analgesia techniques in pediatric/adolescent patients undergoing orthopedic procedures, particularly ambulatory knee procedures such as anterior cruciate ligament (ACL) reconstruction and medial patellofemoral ligament (MPFL) reconstruction. Given the innervation to the knee and concern with residual functional impairment, the goal of our pilot study is to collect preliminary information comparing the anterior femoral cutaneous nerve block (AFCNB) vs adductor canal block (ACB), in the hopes of using this data to power a larger randomized controlled trial to rigorously study this clinical question.

This pilot clinical trial aims to find out what the differences are between anterior femoral cutaneous nerve block (AFCN) and adductor canal block (ACB) for pediatric patients who are having either anterior cruciate ligament (ACL) or medial patellofemoral ligament (MPFL) surgery. There will be 30 subjects in each group/type of surgery. The aims of this trial are:

* To measure postoperative functional outcomes in patients who received AFCNB vs. ACB.
* To calculate postoperative opioid requirements in pediatric knee surgeries that received AFCNB vs. ACB.
* To calculate pain intensity levels at rest and with ambulation in patients who received AFCNB vs. ACB.
* To quantify sensory deficits in patients who received AFCNB vs. ACB.
* To assess patient-reported outcome measures (e.g., pain expectation scale, pain management satisfaction, PROMIS Pediatric Short Form v1.0 - Physical Activity, PROMIS Scale v1.2 - Global Health) in patients 8-18 years of age who received AFCNB vs. ACB.

  30 Subjects undergoing ACL procedures will be compared between those who received the adductor canal block (15) to those who received the anterior femoral cutaneous nerve block (15). The researchers will also compare 30 individuals who underwent MPFL procedures and received an anterior femoral cutaneous nerve block (15) with those who received the adductor canal block (15).

Eligible and enrolled participants will:

* Be randomized to receive either the AFCNB or ACB in addition to standard of care analgesia.
* Maintain a patient diary to document daily pain meds/pain scores
* Complete follow up surveys/questionnaires via telephone and during their office visits with surgeons.

ELIGIBILITY:
Inclusion Criteria:

* 8-18 years old at the time of surgery
* Patients 40kg and above
* ACL reconstruction of MPFL reconstruction surgery with participating surgeons

Exclusion Criteria:

* revision surgery
* bilateral surgery
* general anesthesia
* contraindications to any part of the study protocol
* relevant pre-existing neurological deficit
* chronic pain

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Function (Motor strength in quadriceps) | 3 months
  Collected at standard of care postoperative clinical visits with surgeon. Quadriceps strength is measured bilaterally by a handheld dynamometer.

SECONDARY OUTCOMES:
Cumulative opioid consumption (MMEs) | 48 hours after surgery
  Opioids administered to or consumed by patient in the first 48 hours after surgery (starting from "PACU in" time to 48 hours after "PACU in" time)
Total opioid consumption (MMEs) | at postoperative day 7 & 14
  defined as cumulative opioid consumption (in MME) from PACU transfer in time to 7 days postoperatively and from PACU transfer in time to 14 days postoperatively
Opioid consumption | at 6 weeks, 3 months, 6 months
  defined as any opioid consumption at 6 weeks, 3 months, 6 months postoperatively
Pain Numerical Rating Scale (NRS) at rest | preop (baseline); every 30 minutes beginning from PACU transfer in time to discharge; at 6 hours, 24 hours, 48 hours, 7 days, 14 days, 6 weeks, 3 months, 6 months postoperatively
  Defined on a scale of 0-10, where 0 is no pain and 10 is the worst pain imaginable.
Pain Numerical Rating Scale (NRS) with ambulation | preop (baseline); in PACU; at 6 hours, 24 hours, 48 hours, 7 days, 14 days, 6 weeks, 3 months, 6 months postoperatively
  Defined on a scale of 0 to 10, where 0 is no pain and 10 is the worst pain imaginable.
Postoperative pain location(s) | at 2 weeks, 6 weeks, 3 months, 6 months
  Collected at standard of care postoperative clinical visits (2 weeks, 6 weeks, 3 months, 6 months). Will be collected on a knee dermatomal map (with incisions depicted) with location(s) of pain marked and average pain scores at each location
Pain expectation scale | at postoperative days 1, 2, 7, and 14
  patient reported on a scale of less, same, or more [or unknown] than expected. With "less" being the lower score and "more" being the higher score.
Satisfaction with pain management | at postoperative days 1, 2, 7, and 14
  measured on a scale from 0 to 10, where 0 is very dissatisfied and 10 is very satisfied with the pain management regimen.
postoperative sensation | at 2 weeks, 6 weeks, 3 months, and 6 months
  collected at standard of care postoperative clinical visits (2 weeks, 6 weeks, 6 months). Will be measured on a knee dermatomal map (with incisions depicted) and classified as "normal," "decreased," or "paresthesia" when compared to the contralateral knee.
postoperative function - motor strength in quadriceps | at 2 weeks, 6 weeks, 6 months
  collected at standard of care postoperative clinical visits with surgeon; quadriceps strength: measured bilaterally by handheld dynamometer
postoperative function - range of motion (ROM) | at 2 weeks, 6 weeks, 3 months, 6 months
  collected at standard of care postoperative clinical visits with surgeon; range of motion (ROM): measured bilaterally by goniometer
postoperative function - Patient-Reported Outcomes Measurement Information System (PROMIS) physical function. | at 2 weeks, 6 weeks, 3 months, 6 months
  collected at standard of care postoperative clinical visits with surgeon; physical function: PROMIS. If the patient is less than 18 years of age, will be assessed using the PROMIS Pediatric Short Form v1.0 - Physical Activity, which contains questions regarding performance of activities such as exercise and play in the past 7 days with 5 answer choices: no days, 1 day, 2-3 days, 4-5 days, and 6-7 days. If the patient is 18 years of age, will be assessed using the PROMIS Scale v1.2 - Global Health, which contains questions regarding physical and mental health rated 1-5, where 1 is worst and 5 is best (physical raw, T, and health scores will be calculated).

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn DelPizzo, MD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu SS, Strodtbeck WM, Richman JM, Wu CL. A comparison of regional versus general anesthesia for ambulatory anesthesia: a meta-analysis of randomized controlled trials. Anesth Analg. 2005 Dec;101(6):1634-1642. doi: 10.1213/01.ANE.0000180829.70036.4F. PMID 16301234
- [Background] Wang C, Liu LD, Bai X. Bibliometric and Visual Analysis of the Current Status and Trends of Postoperative Pain in Children from 1950-2021. J Pain Res. 2022 Oct 14;15:3209-3222. doi: 10.2147/JPR.S380842. eCollection 2022. PMID 36267350
- [Background] Micalizzi RA, Williams LA, Pignataro S, Sethna NF, Zurakowski D. Review of outcomes in pediatric patients undergoing anterior cruciate ligament repairs with regional nerve blocks. J Pediatr Nurs. 2014 Nov-Dec;29(6):670-8. doi: 10.1016/j.pedn.2014.07.002. Epub 2014 Jul 13. PMID 25089833
- [Background] Walker BJ, Long JB, Sathyamoorthy M, Birstler J, Wolf C, Bosenberg AT, Flack SH, Krane EJ, Sethna NF, Suresh S, Taenzer AH, Polaner DM, Martin L, Anderson C, Sunder R, Adams T, Martin L, Pankovich M, Sawardekar A, Birmingham P, Marcelino R, Ramarmurthi RJ, Szmuk P, Ungar GK, Lozano S, Boretsky K, Jain R, Matuszczak M, Petersen TR, Dillow J, Power R, Nguyen K, Lee BH, Chan L, Pineda J, Hutchins J, Mendoza K, Spisak K, Shah A, DelPizzo K, Dong N, Yalamanchili V, Venable C, Williams CA, Chaudahari R, Ohkawa S, Usljebrka H, Bhalla T, Vanzillotta PP, Apiliogullari S, Franklin AD, Ando A, Pestieau SR, Wright C, Rosenbloom J, Anderson T; Pediatric Regional Anesthesia Network Investigators. Complications in Pediatric Regional Anesthesia: An Analysis of More than 100,000 Blocks from the Pediatric Regional Anesthesia Network. Anesthesiology. 2018 Oct;129(4):721-732. doi: 10.1097/ALN.0000000000002372. PMID 30074928
- [Background] Yee EJ, Gapinski ZA, Ziemba-Davis M, Nielson M, Meneghini RM. Quadriceps Weakness After Single-Shot Adductor Canal Block: A Multivariate Analysis of 1,083 Primary Total Knee Arthroplasties. J Bone Joint Surg Am. 2021 Jan 6;103(1):30-36. doi: 10.2106/JBJS.19.01425. PMID 33079899
- [Background] Zhao XQ, Jiang N, Yuan FF, Wang L, Yu B. The comparison of adductor canal block with femoral nerve block following total knee arthroplasty: a systematic review with meta-analysis. J Anesth. 2016 Oct;30(5):745-54. doi: 10.1007/s00540-016-2194-1. Epub 2016 Jun 4. PMID 27262287
- [Background] Kuang MJ, Ma JX, Fu L, He WW, Zhao J, Ma XL. Is Adductor Canal Block Better Than Femoral Nerve Block in Primary Total Knee Arthroplasty? A GRADE Analysis of the Evidence Through a Systematic Review and Meta-Analysis. J Arthroplasty. 2017 Oct;32(10):3238-3248.e3. doi: 10.1016/j.arth.2017.05.015. Epub 2017 May 17. PMID 28606458
- [Background] Jiang X, Wang QQ, Wu CA, Tian W. Analgesic Efficacy of Adductor Canal Block in Total Knee Arthroplasty: A Meta-analysis and Systematic Review. Orthop Surg. 2016 Aug;8(3):294-300. doi: 10.1111/os.12268. PMID 27627711
- [Background] Abdallah FW, Brull R, Joshi GP; Society for Ambulatory Anesthesia (SAMBA). Pain Management for Ambulatory Arthroscopic Anterior Cruciate Ligament Reconstruction: Evidence-Based Recommendations From the Society for Ambulatory Anesthesia. Anesth Analg. 2019 Apr;128(4):631-640. doi: 10.1213/ANE.0000000000003976. PMID 30649069
- [Background] Abdallah FW, Whelan DB, Chan VW, Prasad GA, Endersby RV, Theodoropolous J, Oldfield S, Oh J, Brull R. Adductor Canal Block Provides Noninferior Analgesia and Superior Quadriceps Strength Compared with Femoral Nerve Block in Anterior Cruciate Ligament Reconstruction. Anesthesiology. 2016 May;124(5):1053-64. doi: 10.1097/ALN.0000000000001045. PMID 26938989
- [Background] Christensen JE, Taylor NE, Hetzel SJ, Shepler JA, Scerpella TA. Isokinetic Strength Deficit 6 Months After Adductor Canal Blockade for Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2017 Nov 8;5(11):2325967117736249. doi: 10.1177/2325967117736249. eCollection 2017 Nov. PMID 29152521
- [Background] Frazer AR, Chausse ME, Held M, St-Pierre C, Tsai CY, Preuss R, Descoteaux N, Chan M, Martineau PA, Veilleux LN. Quadriceps and Hamstring Strength in Adolescents 6 Months After ACL Reconstruction With Femoral Nerve Block, Adductor Canal Block, or No Nerve Block. Orthop J Sports Med. 2021 Jul 22;9(7):23259671211017516. doi: 10.1177/23259671211017516. eCollection 2021 Jul. PMID 34368383
- See also: Anterior Femoral Cutaneous Nerve Block (Dr. Jeff Gadsden) — http://www.youtube.com/watch?v=zzj08axeE94
- See also: Anterior Femoral Cutaneous Nerve Block (Dr. Amit Pawa) — http://www.youtube.com/watch?v=bAxMvcTf0kU

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT06590402/Prot_SAP_000.pdf